CLINICAL TRIAL: NCT01493505
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study of AMG 386 With Paclitaxel and Carboplatin as First-line Treatment of Subjects With FIGO Stage III-IV Epithelial Ovarian, Primary Peritoneal or Fallopian Tube Cancers
Brief Title: TRINOVA-3: A Study of AMG 386 or AMG 386 Placebo in Combination With Paclitaxel and Carboplatin to Treat Ovarian Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Amgen Administrative Decision - termination of LTFU
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20101129; TRINOVA-3 20101129/ENGOT-ov2
Record Dates: First submitted 2011-09-29; First posted 2011-12-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cancer
Keywords: Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — trebananib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo Paclitaxel Carboplatin
  Interventions: Drug: Paclitaxel; Drug: AMG 386 Placebo; Drug: Carboplatin
- AMG 386 (Active Comparator): AMG 386 Paclitaxel Carboplatin
  Interventions: Drug: AMG 386; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: AMG 386 — AMG 386 15mg/kg IV QW (until progression or unacceptable toxicity develops)
  Arms: AMG 386
Drug: Paclitaxel — Paclitaxel 175 mg/m2 3 hour IV Q3W (6 cycles)
Drug: AMG 386 Placebo — AMG 386 Placebo IV QW (until progression or unacceptable toxicity develops)
  Arms: Placebo
Drug: Carboplatin — Carboplatin AUC 5 or 6 IV Q3W (6 cycles)

SUMMARY:
The purpose of this study is to determine whether AMG 386 or AMG 386 Placebo in combination with Paclitaxel and Carboplatin are effective in the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 18 years of age or older with FIGO Stages III-IV epithelial ovarian, primary peritoneal or fallopian tube cancer with an indication for first-line treatment with paclitaxel and carboplatin x 6 cycles (Subjects with pseudomyxoma, mesothelioma, adenocarcinoma with an unknown primary tumour, carcinosarcoma, sarcoma, mucinous or neuroendocrine histology are excluded
* Subjects with FIGO Stage IIIA or IIIB disease must have undergone PDS for ovarian, primary peritoneal or fallopian tube cancer within 12 weeks prior to randomization
* Subjects with FIGO Stage IIIC or IV disease must either:
* Undergo PDS for epithelial ovarian, primary peritoneal or fallopian tube cancer within 12 weeks prior to randomization or
* Plan to have IDS following 3 cycles of paclitaxel and carboplatin plus AMG 386 or AMG 386 placebo for biopsy proven epithelial ovarian, primary peritoneal or fallopian tube cancer
* ECOG performance status of 0 or 1
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Prior use of any anticancer therapy or experimental therapy for epithelial ovarian, primary peritoneal or fallopian tube cancer
* Previous abdominal and/or pelvic external beam radiotherapy
* History of central nervous metastasis
* History of arterial or venous thromboembolism within 12 months prior to randomization
* Clinically significant cardiovascular disease within 12 months prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
Incidence of adverse events and significant laboratory abnormalities | 4 years
Pharmacokinetics of AMG 386 (Cmax and Cmin) | 1 year
  pre-dose weeks 1, 7, 10, 19 and within 10 minutes post dose week 1, 7
Incidence of anti-AMG 386 antibody formation | 4 years
  pre-dose weeks 1, 10, 19
Patient reported ovarian cancer-specific symptoms and health related quality of life | 4 years
Patient reported status as measured by the EuroQOL (EQ-5D) | 4 years
AMG 386 exposure-response relationships for PFS and OS | 4 years
Correlation of serum biomarkers with measures of response | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (256):
- United States (145):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Gilbert, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Berkeley, California
  - Research Site, Burbank, California
  - Research Site, Concord, California
  - Research Site, Corona, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Oxnard, California
  - Research Site, Rancho Mirage, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Aurora, Colorado
  - Research Site, Englewood, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Farmington, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, New Britain, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Ames, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Edgewood, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Danvers, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Research Site, Neptune City, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Brightwaters, New York
  - Research Site, Buffalo, New York
  - Research Site, Jamaica, New York
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Concord, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Mayfield Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Radnor, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Ogden, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Annandale, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Woodbridge, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, Marshfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Oshkosh, Wisconsin
  - Research Site, Sheboygan, Wisconsin
  - Research Site, Waukesha, Wisconsin
  - Research Site, Wausau, Wisconsin
  - Research Site, West Allis, Wisconsin
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (18):
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Duffel
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Libramont
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Sint-Niklaas
  - Research Site, Turnhout
  - Research Site, Wilrijk
  - Research Site, Yvoir
- Canada (9):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (3):
  - Research Site, Herlev
  - Research Site, København Ø
  - Research Site, Roskilde
- Germany (20):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Kiel
  - Research Site, Konstanz
  - Research Site, Leipzig
  - Research Site, Ludwigsburg
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Ravensburg
  - Research Site, Rostock
  - Research Site, Stuttgart
  - Research Site, Tübingen
  - Research Site, Ulm
- Greece (4):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Kowloon
  - Research Site, New Territories
- Italy (13):
  - Research Site, Avellino
  - Research Site, Aviano PN
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Japan (11):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kashiwa, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Kure, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Morioka, Iwate
  - Research Site, Kitaadachi-gun, Saitama
  - Research Site, Suntou-gun, Shizuoka
  - Research Site, Yonago, Tottori
  - Research Site, Tokyo
- Netherlands (4):
  - Research Site, Deventer
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Russia (9):
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Voronezh
- South Korea (2):
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seoul
- Spain (10):
  - Research Site, Zaragoza, Aragon
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Girona, Catalonia
  - Research Site, Lleida, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia

REFERENCES:
- [Background] Fujiwara K, Monk BJ, Lhomme C, Coleman RL, Brize A, Oaknin A, Ray-Coquard I, Fabbro M, Provencher D, Bamias A, Vergote I, DeCensi A, Zhang K, Vogl FD, Bach BA, Raspagliesi F. Health-related quality of life in women with recurrent ovarian cancer receiving paclitaxel plus trebananib or placebo (TRINOVA-1). Ann Oncol. 2016 Jun;27(6):1006-1013. doi: 10.1093/annonc/mdw147. Epub 2016 Mar 30. PMID 27029706
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Vergote I, Scambia G, O'Malley DM, Van Calster B, Park SY, Del Campo JM, Meier W, Bamias A, Colombo N, Wenham RM, Covens A, Marth C, Raza Mirza M, Kroep JR, Ma H, Pickett CA, Monk BJ; TRINOVA-3/ENGOT-ov2/GOG-3001 investigators. Trebananib or placebo plus carboplatin and paclitaxel as first-line treatment for advanced ovarian cancer (TRINOVA-3/ENGOT-ov2/GOG-3001): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2019 Jun;20(6):862-876. doi: 10.1016/S1470-2045(19)30178-0. Epub 2019 May 7. PMID 31076365
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com